CLINICAL TRIAL: NCT02611895
Title: Testing the Effect of Raltegravir on Persistent de Novo HIV Infection in Virologic Responders to Antiretroviral Therapy ( RALNOVO )
Brief Title: Testing the Effect of Raltegravir on Persistent de Novo HIV Infection in Virologic Responders to Antiretroviral Therapy
Acronym: RALNOVO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Institute of Human Genetics, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9503
Record Dates: First submitted 2015-11-19; First posted 2015-11-23 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: HIV-1 Infection
Keywords: Aviremic HIV-1 infected patients; HAART; Integrase inhibitor Raltegravir; Ongoing HIV infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HIV DNA (Experimental): Blood test : Quantitate the amount of HIV DNA harbored in the cytoplasm of peripheral blood CD4+ T cells
  Interventions: Biological: HIV DNA

INTERVENTIONS:
Biological: HIV DNA — Quantitate the amount of HIV DNA harbored in the cytoplasm of peripheral blood CD4+ T cells

SUMMARY:
There is a theoretical possibility of a complete suppression of HIV viral replication, subject to the use of highly active associations of more than 25 antiretroviral drugs currently available and good treatment adherence. But a key question remains: whether it can persist viral replication low noise HAART, since several arguments suggest a subclinical escape of the virus to HAART at least in some individuals. The technique proposed in this research consists of the detection and quantification of the linear viral cDNA intra cytoplasmic, as persistent novo infection marker in order to highlight the subclinical replication active in treatment of HIV-1 and consider an optimized therapeutic management of patients.

Main objective : Comparing the frequency of patients infected with HIV and treated effectively (HIV viral load undetectable plasma with conventional methods) having the HIV DNA into the cytoplasm of their CD4 + T cells from peripheral blood, as cellular infection marker novo persistent, among patients with a therapeutic regimen contains or not the viral integrase inhibitor raltegravir.

Secondary objectives

* To evaluate the frequency of patients infected with HIV and treated effectively with the HIV DNA into the cytoplasm of their CD4 + T cells from peripheral blood
* Evaluate the causes of persistent infection in de novo virological responders to treatment with ART: presence of the HIV genome encoding strains resistant to treatment ART ongoing noncompliance to treatment, type of antiretroviral therapy, CD4 nadir , pretreatment level of plasma HIV RNA, total duration of ART
* Assess the impact of persistent novo infection virological responders: cell activation CD4 + and CD8 +, lack of immunological treatment response, changes in lymphocyte ratio T naïve / memory cells cells, the presence of transient increase viremia, residual viremia levels
* Identify virological responders may benefit from treatment intensification

DETAILED DESCRIPTION:
There is a theoretical possibility of a complete suppression of HIV viral replication, subject to the use of highly active associations of more than 25 antiretroviral drugs currently available and good treatment adherence. But a key question remains: whether it can persist viral replication low noise HAART, since several arguments suggest a subclinical escape of the virus to HAART at least in some individuals. The technique proposed in this research consists of the detection and quantification of the linear viral cDNA intra cytoplasmic, as persistent novo infection marker in order to highlight the subclinical replication active in treatment of HIV-1 and consider an optimized therapeutic management of patients.

Main objective : Comparing the frequency of patients infected with HIV and treated effectively (HIV viral load undetectable plasma with conventional methods) having the HIV DNA into the cytoplasm of their CD4 + T cells from peripheral blood, as cellular infection marker novo persistent, among patients with a therapeutic regimen contains or not the viral integrase inhibitor raltegravir.

Secondary objectives

* To evaluate the frequency of patients infected with HIV and treated effectively with the HIV DNA into the cytoplasm of their CD4 + T cells from peripheral blood
* Evaluate the causes of persistent infection in de novo virological responders to treatment with ART: presence of the HIV genome encoding strains resistant to treatment ART ongoing noncompliance to treatment, type of antiretroviral therapy, CD4 nadir , pretreatment level of plasma HIV RNA, total duration of ART
* Assess the impact of persistent novo infection virological responders: cell activation CD4 + and CD8 +, lack of immunological treatment response, changes in lymphocyte ratio T naïve / memory cells cells, the presence of transient increase viremia, residual viremia levels
* Identify virological responders may benefit from treatment intensification Methods : HIV patients will be recruited by the doctors of Infectious and Tropical Diseases Service (MIT) in the Montpellier University Hospital.

As part of this research, three additional blood tubes (7 ml EDTA tube) will be collected, totaling 21 ml at the time of blood sampling carried out during two consultations scheduled as part of the usual care the pathology of HIV patients in the Service of MIT.

These consultations will be conducted at baseline and a further 3 to 6 months from the date of inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years
* HIV-1 infection
* Current number of T CD4+ lymphocytes > 200 cells / mm3 for 6 moths before inclusion
* Efficient and well tolerated antiretroviral treatment for more than 12 months
* HIV-1 viral load < 50 copies/ml for more than 12 months before inclusion
* Patient able to understand the nature, the objective and the methods of the study
* Patient having signed the informed consent
* Affiliation to French Social Security System

Exclusion Criteria:

* Patient is currently participating or has participated in a study (within the exclusion period defined by this study)
* Patient is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-03-22 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Frequency of virologic responders harbouring intracytoplasmic HIV DNA in their peripheral blood CD4+ T cells, used as a surrogate marker of ongoing HIV infection, between subjects whose regimen contains or not the integrase inhibitor raltegravir. | 1 day
  Frequency of virologic responders harbouring intracytoplasmic HIV DNA in their peripheral blood CD4+ T cells, used as a surrogate marker of ongoing HIV infection, between subjects whose regimen contains or not the integrase inhibitor raltegravir.

SECONDARY OUTCOMES:
Causes and consequences of persistent de novo infection in virologic responders to HAART | 1 day
  Causes and consequences of persistent de novo infection in virologic responders to HAART

CONTACTS AND LOCATIONS:
Overall Officials: CHRISTINA PSOMAS, Principal Investigator — University Hospital of Montpellier, Montpellier, France, 34295
Locations (1):
- University hospital Montpellier, Montpellier, France